CLINICAL TRIAL: NCT05505916
Title: An Open-label Extension Trial to Evaluate the Long-term Safety of KVD900, an Oral Plasma Kallikrein Inhibitor, for On-demand Treatment of Angioedema Attacks in Adolescent and Adult Patients With Hereditary Angioedema Type I or II
Brief Title: An Open-label Extension Trial to Evaluate the Long-term Safety of KVD900 (Sebetralstat) for On-Demand Treatment of Angioedema Attacks in Adolescent and Adult Patients With Hereditary Angioedema (HAE)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KVD900-302
Record Dates: First submitted 2022-08-11; First posted 2022-08-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hereditary Angioedema
Keywords: KONFIDENT-S; Sebetralstat
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — sebetralstat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KVD900 600 mg (Experimental)
  Interventions: Drug: KVD900 600 mg
- KVD900 300 mg (Experimental)
  Interventions: Drug: KVD900 300 mg

INTERVENTIONS:
Drug: KVD900 600 mg — KVD900 Tablet 600 mg (2 x 300 mg)
  Arms: KVD900 600 mg
Drug: KVD900 300 mg — KVD900 Tablet 300 mg
  Arms: KVD900 300 mg

SUMMARY:
This is an open-label, multicenter extension trial to evaluate the long-term safety of KVD900 in patients who are 12 years or older with HAE type I or II.

ELIGIBILITY:
Patients may roll over from KVD900-301.

Inclusion Criteria:

1. Confirmed diagnosis of HAE type I or II at any time in the medical history
2. Patient has had at least 2 documented HAE attacks within 3 months prior to the Enrollment Visit.
3. If a patient is receiving long-term prophylactic treatment with one of the protocol-allowed therapies, they must have been on a stable dose and regimen for at least 3 months prior to the Enrollment Visit (except for danazol, which requires a stable dose and regimen for at least 6 months prior to the Enrollment Visit).
4. Male or female patients 12 years of age and older.
5. Patients must meet the contraception requirements.
6. Patients must be able to swallow trial tablets whole.
7. Patients, as assessed by the Investigator, must be able to appropriately receive and store IMP, and be able to read, understand, and complete the eDiary.
8. Investigator believes that the patient is willing and able to adhere to all protocol requirements.
9. Patient provides signed informed consent or assent (when applicable). A parent or legally authorized representative (LAR) must also provide signed informed consent when required.

Exclusion Criteria:

1. Discontinued from the KVD900-301 trial for reasons of noncompliance, withdrawal of consent, or safety.
2. Presence of any safety concerns that would preclude participation in the open-label trial as determined by the investigator.
3. Any concomitant diagnosis of another form of chronic angioedema, such as acquired C1 inhibitor deficiency, HAE with normal C1-INH (previously known as HAE type III), idiopathic angioedema, or angioedema associated with urticaria.
4. A clinically significant history of poor response to bradykinin receptor 2 (BR2) blocker, C1-INH therapy, or plasma kallikrein inhibitor therapy for the management of HAE, in the opinion of the Investigator.
5. Use of attenuated androgens other than danazol (e.g., stanozolol, oxandrolone, methyltestosterone, testosterone), or anti-fibrinolytics (e.g., tranexamicacid) within 28 days prior to the Enrollment Visit.
6. Use of Angiotensin-converting enzyme (ACE) inhibitors within 7 days prior to the Enrollment Visit.
7. Any estrogen-containing medications with systemic absorption (such as oral contraceptives including ethinylestradiol or hormonal replacement therapy) within 7 days prior to the Enrollment Visit.
8. Inadequate organ function, including but not limited to:

   1. Alanine aminotransferase (ALT) >2x Upper Limit Normal (ULN)
   2. Aspartate aminotransferase (AST) >2x ULN
   3. Bilirubin direct >1.25x ULN
   4. International Normalized Ratio (INR) >1.2
   5. Clinically significant hepatic impairment defined as a Child-Pugh B or C
9. Any clinically significant comorbidity or systemic dysfunction, which in the opinion of the Investigator, would jeopardize the safety of the patient by participating in the trial.
10. History of substance abuse or dependence that would interfere with the completion of the trial, as determined by the Investigator.
11. Known hypersensitivity to KVD900 or to any of the excipients.
12. Participation in any gene therapy treatment or trial for HAE.
13. Participation in any interventional investigational clinical trial, including an investigational COVID-19 vaccine trial, within 4 weeks of the last dosing of investigational drug prior to the Enrollment Visit.
14. Any pregnant or breastfeeding patient.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequencies and percentages of patients with AEs, AEs within 2 days of IMP administration, serious AE's and AEs causing premature discontinuation. | AEs will be recorded from the first dose of IMP in the KVD900-302 trial up to and including the end of study (EOS) visit, a maximum of 2 years for each patient.
Number and percentage of patients with normal or abnormal laboratory results at each scheduled visit. | Throughout the duration of the trial.
Number and percentage of patients with normal or abnormal vital sign results at each scheduled visit | Throughout the duration of the trial.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGI-C). | within 12 hours of initial dose of IMP administration.
  time to beginning of symptom relief defined as at least '' a little better'' (2 time points in a row)
Patient Global Impression of Severity (PGI-S): time to first incidence of 2 time points in a row decrease from baseline | within 12 hours of initial dose of IMP administration.
PGI-S: time to HAE attack resolution | within 24 hours of initial dose of IMP administration.
  PGI-S: time to HAE attack resolution, defines as ''none''

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — KalVista Pharmaceuticals, Ltd.
Locations (67):
- United States (19):
  - KalVista Investigative Site, Scottsdale, Arizona
  - KalVista Investigative Site, Little Rock, Arkansas
  - KalVista Investigative Site, San Diego, California
  - KalVista Investigative Site, Santa Monica, California
  - KalVista Investigative Site, Centennial, Colorado
  - KalVista Investigative Site, Colorado Springs, Colorado
  - KalVista Investigative Site, Evansville, Indiana
  - KalVista Investigative Site, Overland Park, Kansas
  - KalVista Investigative Site, Louisville, Kentucky
  - KalVista Investigative Site, Chevy Chase, Maryland
  - KalVista Investigative Site, Plymouth, Minnesota
  - KalVista Investigative Site, St Louis, Missouri
  - KalVista Investigative Site, Charlotte, North Carolina
  - KalVista Investigative Site, Cincinnati, Ohio
  - KalVista Investigative Site, Toledo, Ohio
  - KalVista Investigative Site, Hershey, Pennsylvania
  - KalVista Investigative Site, Dallas, Texas
  - KalVista Investgative Site, Layton, Utah
  - KalVista Investigative Site, Spokane, Washington
- KalVista Investigative Site, Campbelltown, Australia
- KalVista Investigative Site, Wein, Austria
- KalVista Investigative Site, Sofia, Bulgaria
- KalVista Investigative Site, Montreal, Canada
- France (3):
  - KalVista Investigative Site, Grenoble
  - KalVista Investigative Site, Lille
  - KalVista Investigative Site, Paris
- Germany (4):
  - KalVista Investigative Site, Berlin
  - KalVista Investigative Site, Frankfurt
  - KalVista Investigative Site, Mainz
  - KalVista Investigative Site, Mörfelden-Walldorf
- KalVista Investigative Site, Athens, Greece
- KalVista Investigative Site, Budapest, Hungary
- Israel (4):
  - KalVista Investigative Site, Haifa
  - KalVista Investigative Site, Petach Tikvah
  - KalVista Investigative Site, Ramat Gan
  - KalVista Investigative Site, Tel Aviv
- Italy (4):
  - KalVista Investigative Site, Padua
  - KalVista Investigative Site, Palermo
  - KalVista Investigative Site, Roma
  - KalVista Investigative Site, San Donato Milanese
- Japan (9):
  - KalVista Investigative Site, Sapporo, Hokkaido
  - KalVista Investigative Site, Chiba
  - KalVista Investigative Site, Hiroshima
  - KalVista Investigative Site, Kawagoe-shi
  - KalVista Investigative Site, Maebashi
  - KalVista Investigative Site, Soka-shi
  - KalVista Investigative Site, Takatsuki-shi
  - KalVista Investgative Site, Tokyo
  - KalVista Investigative Site, Yokohama
- KalVista Investigative Site, Amsterdam, Netherlands
- KalVista Investigative Site, Auckland, New Zealand
- KalVista Investigative Site, Skopje, North Macedonia
- Poland (2):
  - KalVista Investigative Site, Krakow
  - KalVista Investigative Site, Lodz
- KalVista Investigative Site, Porto, Portugal
- KalVista Investigative Site, Sângeorgiu de Mureş, Romania
- KalVista Investigative Site, Riyadh, Saudi Arabia
- KalVista Investigative Site, Martin, Slovakia
- Kalvista Investigative Site, Cape Town, South Africa
- Spain (2):
  - KalVista Investigative Site, Barcelona
  - KalVista Investigative Site, Madrid
- United Kingdom (6):
  - KalVista Investigative Site, Birmingham
  - KalVista Investigative Site, Cambridge
  - KalVista Investigative Site, Cardiff
  - KalVista Investigative Site, Frimley
  - KalVista Investigative Site, Leeds
  - KalVista Investigative Site, London

IPD SHARING:
Plan to Share IPD: No
Data will not be shared until all global regulatory filings are complete.

REFERENCES:
- [Derived] Bernstein JA, Aygoren-Pursun E, Cancian M, Cohn DM, Craig T, Grivcheva-Panovska V, Jordan A, Lumry WR, Martinez-Saguer I, Melamed I, Ohmura K, Peter J, Riedl MA, Soteres DF, Staubach P, Stobiecki M, Chuang YH, Smith MD, Yea CM, Audhya PK, Zanichelli A, Farkas H. Sebetralstat for On-Demand Treatment of Mucosal Hereditary Angioedema Attacks in KONFIDENT-S. Clin Transl Allergy. 2025 Nov;15(11):e70118. doi: 10.1002/clt2.70118. PMID 41252457
- [Derived] Farkas H, Anderson J, Bouillet L, Caballero T, Cancian M, Craig T, Fukunaga A, Grivcheva-Panovska V, Guilarte M, Honda D, Kanarek H, Kiani-Alikhan S, Kinaciyan T, Leguevaques D, Longhurst HJ, Magerl M, Manning ME, Martinez-Saguer I, Melamed I, O'Connor ME, Peter J, Savic S, Soteres DF, Staevska M, Staubach P, Stobiecki M, Tachdjian R, Valerieva A, Yong PFK, Hao J, Iverson M, Smith MD, Yea CM, Audhya PK, Aygoren-Pursun E, Bernstein JA, Cohn DM, Lumry WR, Riedl MA, Zanichelli A, Maurer M. Long-Term Safety and Effectiveness of Sebetralstat: Interim Analysis of KONFIDENT-S Open-label Extension. J Allergy Clin Immunol Pract. 2025 Nov;13(11):3094-3103.e5. doi: 10.1016/j.jaip.2025.08.020. Epub 2025 Aug 29. PMID 40886933